CLINICAL TRIAL: NCT01892839
Title: Increasing the Removal of Protein-Bound Solutes During Extended Hours Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MEY0026APR
Record Dates: First submitted 2013-06-27; First posted 2013-07-04 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: End Stage Renal Failure on Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high dialysate flow, larger dialyzer (Experimental): high dialysate flow, larger dialyzer
  Interventions: Other: high dialysate flow, larger dialyzer
- low dialysate flow, smaller dialyzer (Active Comparator): low dialysate flow, smaller dialyzer
  Interventions: Other: low dialysate flow, smaller dialyzer

INTERVENTIONS:
Other: low dialysate flow, smaller dialyzer — The subject will receive dialysis on the usual schedule and for the usual time but with a lower than usual dialysate flow and small dialyzer.
  Arms: low dialysate flow, smaller dialyzer
Other: high dialysate flow, larger dialyzer — The subject will receive dialysis on the usual schedule and for the usual time but with a higher than usual dialysate flow and large dialyzer.
  Arms: high dialysate flow, larger dialyzer

SUMMARY:
Hemodialysis keeps patients with renal failure alive but does not restore normal health. Retention of chemicals that bind to plasma proteins and are therefore poorly removed by dialysis may contribute to ill health in patients receiving conventional treatment. This proposal will test the effect of a new method designed to improve the removal of protein-bound solutes during dialysis. The effects on blood chemical levels of two different dialysis prescriptions will be tested in patients already undergoing nocturnal in-center hemodialysis three times weekly.

ELIGIBILITY:
Inclusion Criteria:

* stable on nocturnal in-center dialysis located close to Stanford University and VA Palo Alto

Exclusion Criteria:

* recent use of antibiotics
* gastrointestinal disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of the chemical p-cresol sulfate | Participants will be followed for 2-3 weeks on different dialysis prescriptions and plasma chemical levels will be measured at the end of this period.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy W Meyer, MD, Principal Investigator — PAIRE
Locations (2):
- United States (2):
  - Satellite Redwood City, Redwood City, California
  - Stanford University, Stanford, California